CLINICAL TRIAL: NCT04246359
Title: Safety and Activity of Rituximab(HLX01) in Combination With Pegylated Interferon α-2b in Patients With Newly Diagnosed Advanced Indolent B-cell Lymphoma: a Single-arm, Multicenter, Phase 2 Study
Brief Title: Rituximab and Pegylated Interferon α-2b in Patients With Indolent B-cell Lymphoma
Acronym: RIPPLE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huiqiang Huang (Other)
Responsible Party: Sponsor-Investigator, Huiqiang Huang, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIPPLE
Record Dates: First submitted 2020-01-14; First posted 2020-01-29 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Lymphoma, B-Cell
Keywords: indolent B-cell lymphoma; Rituximab(HLX01); Pegylated Interferon α-2b; HBsAg clearance rate
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RP induction and maintenance (Experimental): 1. Induction phase:
  1. Rituximab: 375mg / m2, ivd, d1;
  2. Pegylated interferon α-2b: 135 μg (500,000 U), H, d1, 8 Repeated every 21 days, Maximum 6 cycles 2. Maintenance phase:
  1) Rituximab: 375mg / m2, ivd, d1; 2) Pegylated interferon α-2b: 135 μg (500,000 U), H, d1,30 Repeated every 2 months, Maximum 12 cycles
  Interventions: Drug: Rituximab Biosimilar; Drug: Pegylated Interferon α-2b

INTERVENTIONS:
Drug: Rituximab Biosimilar — To evaluate the short-term objective efficacy of HLX01 combined with Pegylated Interferon α-2b in patients with advanced idolent B-cell lymphoma.
  Other Names: HLX01
Drug: Pegylated Interferon α-2b — To evaluate the short-term objective efficacy of HLX01 combined with Pegylated Interferon α-2b in patients with advanced idolent B-cell lymphoma.

SUMMARY:
A phase 2 open label study to evaluate safety and activity of Rituximab(HLX01) in combination with Pegylated interferon α-2b in patients with newly diagnosed advanced indolent B-cell lymphoma.

DETAILED DESCRIPTION:
Indolent B-cell lymphomas (iBCL), including follicular lymphoma (FL), marginal zone lymphoma (MZL), lymphoplasmacytic lymphoma (LPL, including Waldenström macroglobulinemia), and some cases of mantle cell lymphoma (MCL), disproportionally affect older individuals.Treatment options are heterogeneous, varying from watchful waiting to intensive combination therapy. Historically, rituximab based regimens have been used as standard immunochemotherapy for iBCL.Use of immunotherapy for indolent lymphoma had been advocated for many years and several studies reported benefit with interferon (IFN) in combination with chemotherapy or rituximab. The positive rate of HBsAg in B-cell NHL is about 30% in China.Pegylated interferon contribute to convert HBsAg to negative. We aim to evaluate safety and activity of Rituximab(HLX01) in combination with Pegylated interferon α-2b in patients with newly diagnosed advanced iBCL and HBsAg clearance rate of hepatitis B patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age, male or female;
2. Patients with a diagnosis of indolent B-cell non-Hodgkin's lymphoma (iNHL),including following subtypes：follicular lymphoma (grade Ⅰ, Ⅱ), intra-nodal and extra-mucosa-associated lymph Tissue marginal zone lymphoma (MALT), spleen marginal zone B-cell lymphoma, lymph node marginal zone lymphoma(MZL), Lymphocele lymphoma (except macroglobulinemia), small lymphocytic lymphoma(SLL);
3. Treatment naive, and Lugano stage III-IV;
4. Life expectancy at least 12 months;
5. At least one evaluable or measurable disease that meets the Lugano 2014 criteria for malignant lymphoma [Evaluable lesions: 18 fluorodeoxyglucose-positron emission tomography (18FDG/PET) examination showed increased local uptake of lymph nodes or extranodal nodes (higher than liver) and PET and /or Computed Tomography (CT) features consistent with lymphoma features; Measurable lesions: nodular lesions> 15mm in diameter or extranodal lesions> 10mm (if only one measurable lesion has previously received radiotherapy, evidence of radiographic progression after radiotherapy is required), and accompanied by 18FDG increased intake]. It is necessary to exclude cases where there is no measurable lesion and diffuse liver 18FDG uptake is increased;
6. ECOG score 0-2;
7. Organs and bone marrow function normally (within 14 days prior to study drug use, without receiving blood transfusion, granulocyte colony-stimulating factors or other related medical support):

   1. Absolute value of neutrophils ≥1.0 × 109 / L;
   2. Platelets ≥50 × 109 / L;
   3. Hemoglobin ≥8 g / dL;
   4. Serum creatinine ≤ 1.5 times Upper Limit Normal (ULN), or creatinine removal rate ≥40mL / min (estimated according to Cockcroft-Gault formula);
   5. serum total bilirubin ≤ 1.5 times ULN;
   6. Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) ≤ 2.5 times ULN;
   7. Coagulation function: International Normalized Ratio (INR)≤1.5 times ULN; Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT) ≤1.5 times ULN (unless the patient is receiving anticoagulant therapy and PT and APTT are within the expected range at the time of screening);
8. Female patients of childbearing age must have a negative pregnancy test at the time of enrollment and are willing to use reliable contraceptive methods, i.e. barrier methods, oral contraceptives, implant methods, skin contraception, long-acting injection contraceptives, intrauterine devices, or tubal ligation;
9. Sign the informed consent.

Exclusion Criteria:

1. Primary CNS lymphoma or secondary CNS involvement;
2. A history of severe allergic reactions to humanized or murine monoclonal antibodies;
3. Patients have active autoimmune disease that requires systemic treatment in the past two years. (hormonal replacement therapy is not considered as a systemic treatment, such as patients with type 1 diabetes, adrenal function due to hypothyroidism that only requires thyroxine replacement therapy, low or pituitary dysfunction which only requires physiological doses of glucocorticoid replacement therapy); Patients with autoimmune disease without systemic treatment in the past two years can be enrolled;
4. Patients who require systemic glucocorticoid therapy or other immunosuppressive therapy within 14 days before study 【patients are permitted to use topical, ocular, intra-articular, intranasal, and inhaled corticosteroids (with very low systemic absorption), to receive short-term (≤ 7 days) preventive treatment with glucocorticoids (such as contrast agent hypersensitivity) or treatment of non-autoimmune diseases (such as delayed onset of hypersensitivity caused by contact allergen】.Low-dose hormone debulking treatment due to large tumor burden is allowed (prednisone 20mg × 7 days or equivalent dose of other hormones are allowed);
5. Have other malignancies in the past 5 years, except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the breast and carcinoma in situ of the cervix after radical treatment;
6. Within 28 days before study treatment, patients receiving systemic anti-tumor treatments, including chemotherapy, immunotherapy, biotherapy (tumor vaccine, cytokine, or growth factor that controls cancer);
7. Major surgery was performed within 28 days before study treatment, or radiotherapy was performed within the first 90 days;
8. Within 7 days before study treatment, patients receiving anti-cancer Chinese herbal medicine or proprietary Chinese medicine treatment;
9. Live vaccines (excluding influenza attenuated vaccines) within 28 days before study treatment;
10. A history of Human Immunodeficiency Virus (HIV) disease Patients with viral infection and / or acquired immunodeficiency syndrome;
11. Patients with active chronic hepatitis B or active hepatitis C. Patients who are Hepatitis B Surface Antigen (HBsAg) or Hepatitis C Virus (HCV) antibodies positive during the screening period must have the Hepatitis B Virus (HBV) DNA titer test (must not higher than 2500 copies/mL or 1000 I /mL) and HCV RNA test (not to exceed the detection limit of the assay 10,000 copies/mL). Patients can enter the study if there is no treatment require. Patients with carriers of hepatitis B virus, stable hepatitis B after treatment (DNA titers of no more than 2500 copies / mL or 1000 IU / mL), and cured hepatitis C can be enrolled;
12. Any active infection requiring systemic anti-infective treatment within 14 days study treatment;
13. Female patients during pregnancy or lactation;
14. Patients with a history of alcohol or drug abuse;
15. Suffering from uncontrollable comorbidities, including but not limited to symptomatic congestive heart failure, uncontrollable hypertension, unstable angina pectoris, active peptic ulcer or bleeding disorders;
16. A history of interstitial lung disease or non-infectious pneumonia. Patients who previously had drug-induced or radioactive non-infectious pneumonia but were asymptomatic were admitted;
17. Patients with a history of mental illness, inability or restricted ability;
18. On the judgement of the investigator, patient's underlying condition may increase his or her risk when receiving study medications or confuse the occurrence of a toxic reaction and its judgment；
19. Patients of considered by investigators unsuitable for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-06-16 (Estimated); Study Completion 2023-01-16 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR)、Complete Remission Rate (CRR)、Partial Remission Rate (PRR) | Up to 21 weeks
  Short-term effcacy according to Lugano 2014 Malignant Lymphoma Evaluation Criteria
HBsAg clearance rate and anti-Hbs antibody positive rate in patients with chronic hepatitis B at 72 weeks | Up to 72 weeks
  Evaluate HBsAg clearance rate and positive rate of anti-Hbs antibody

SECONDARY OUTCOMES:
Progression Free Survival (PFS) time, | Up to 3 years
  PFS is defined as the time from the treatment date to the date of disease
Duration of Response (DOR) | Up to 3 years
  Evaluate long-term survival time
Overall survival(OS) | Up to 5 years
  Evaluate long-term survival time
Frequency and severity of adverse events (AE), frequency of Serious Adverse Event (SAE) | Up to 2 years
  Incidence and Severity of Toxicities
Ratio of Physical Function and Fatigue Improvement by EORTC Quality of Life Scale QLQ-C30 (V3.0) (on the first day of each course and at each follow-up, up to 60 months) | Up to 2 years
  Quality of Life evaluation to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Ye Cao, Professor, Principal Investigator — Ethics Committee of Cancer Center of Sun Yat-sen University
Locations (1):
- Department of Medical Oncology, Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong, China